CLINICAL TRIAL: NCT05012618
Title: A Phase 1 Open-label, Dose-escalation and Cohort Expansion Study of LUNA18 Monotherapy and Combination Therapy in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Dose-escalation Study of LUNA18 in Patients With Locally Advanced or Metastatic Solid Tumors (With Expansion).
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to discontinue this study upon having LPLV.
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUN101JG
Record Dates: First submitted 2021-08-03; First posted 2021-08-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose escalation part (Part A) (Experimental): Patients will receive LUNA18 capsule(s) at escalated doses
  Interventions: Drug: LUNA18
- Biomarker part (Part B) (Experimental): Patients will receive LUNA18 capsule(s) at doses where the tolerability is confirmed in Part A
  Interventions: Drug: LUNA18
- Cohort expansion part (Part C) (Experimental): Patients will receive LUNA18 capsule(s) at the recommended dose
  Interventions: Drug: LUNA18
- Backfill part (Part AA) (Experimental): Patients will receive LUNA18 capsule(s) at doses where the tolerability is confirmed in Part A
  Interventions: Drug: LUNA18
- Dose finding part (Part D) (Experimental): Patients will receive LUNA18 capsule(s) in combination with cetuximab at finding doses
  Interventions: Drug: LUNA18; Drug: Cetuximab
- Cohort expansion part (Part E) (Experimental): Patients will receive LUNA18 capsule(s) in combination with cetuximab at the recommended dose
  Interventions: Drug: LUNA18; Drug: Cetuximab

INTERVENTIONS:
Drug: LUNA18 — LUNA18 Capsule
Drug: Cetuximab — Cetuximab as a IV infusion
  Arms: Cohort expansion part (Part E); Dose finding part (Part D)

SUMMARY:
This is a Phase 1 dose-escalation and cohort expansion study that will evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary activity of LUNA18 when administered as a single agent or in combination with other anti-cancer drugs in patients with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at time of signing informed consent form
* ECOG performance status of 0 or 1
* Patients with a histologically or cytologically proven diagnosis of a locally advanced, recurrent, or metastatic incurable solid tumor for which standard therapy either does not exist or has proven ineffective or intolerable
* Patients with documented RAS alterations positive solid tumors
* Patients with measurable disease per RECIST v1.1

Exclusion Criteria:

* Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), unstable angina, or myocardial infarction within the previous 6 months or unstable arrhythmias within the previous 3 months
* Patients with primary central nervous system (CNS) malignancy, untreated CNS metastases requiring any anti-tumor treatment, or active CNS metastases
* Patients with current severe, uncontrolled systemic disease (including, but not limited to, clinically significant cardiovascular disease, pulmonary disease, or renal disease, ongoing or active infection)
* Patients with a history or complication of interstitial lung disease (ILD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of LUNA18 (Dose-limiting toxicities) when administered as a single agent [Part A] and in combination with other anti-cancer drugs [Part D] | From Cycle 0 Day 1 until Cycle 1 Day 28 (Cycle 0 is 6-9 days, and Cycle 1 is 28 days)
  Incidence and nature of dose-limiting toxicities (DLTs)
Safety and tolerability of LUNA18 (Adverse Events) [Part A, AA, B, C, D and E] | From Cycle 0 Day 1 (Cycle 0 is 6-9 days) until study completion or treatment discontinuation (up to approximately 43 months)
  Incidence, nature and severity of adverse events, with severity determined per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0)
Plasma concentrations of LUNA18 when administered as a single agent [Part A, AA] and in combination with other anti-cancer drugs [Part D] | From Cycle 0 Day 1 (Cycle 0 is 6-9 days) until study completion or treatment discontinuation (up to approximately 43 months)
  Plasma concentrations of LUNA18
Maximum plasma concentration (Cmax) of LUNA18 when administered as a single agent [Part A, AA] and in combination with other anti-cancer drugs [Part D] | From Cycle 0 Day 1 (Cycle 0 is 6-9 days) until study completion or treatment discontinuation (up to approximately 43 months)
  Maximum plasma concentration (Cmax) of LUNA18
Time to reach maximum plasma drug concentration (Tmax) of LUNA18 when administered as a single agent [Part A, AA] and in combination with other anti-cancer drugs [Part D] | From Cycle 0 Day 1 (Cycle 0 is 6-9 days) until study completion or treatment discontinuation (up to approximately 43 months)
  Time to reach maximum plasma drug concentration (Tmax) of LUNA18
Area under the concentration versus time curve (AUC) of LUNA18 when administered as a single agent [Part A, AA] and in combination with other anti-cancer drugs [Part D] | From Cycle 0 Day 1 (Cycle 0 is 6-9 days) until study completion or treatment discontinuation (up to approximately 43 months)
  Area under the concentration versus time curve (AUC) of LUNA18
Phosphorylation level of ERK protein (pERK) in tumor tissues [Part B] | From screening until the time of clinical responses and/or the time of progressive disease (up to approximately 43 months), if feasible
  Phosphorylation level of ERK protein (pERK) in tumor tissues biomarkers as applicable in tumor tissues
Preliminary anti-tumor activity of LUNA18 when administered as a single agent [Part B, C] and in combination with other anti-cancer drugs [Part E] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first (up to approximately 43 months)
  Objective response, defined as a confirmed complete response (CR) or partial response (PR) as best overall response per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Preliminary anti-tumor activity of LUNA18 when administered as a single agent [Part A, Part AA] and in combination with other anti-cancer drugs [Part D] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first (up to approximately 43 months)
  Objective response, defined as CR or PR as best overall response per RECIST v1.1
Preliminary anti-tumor activity of LUNA18 [Part A, AA, B, C, D and E] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first (up to approximately 43 months)
  Disease control, defined as CR, PR and stable disease (SD) per RECIST v1.1
Preliminary anti-tumor activity of LUNA18 [Part A, AA, B, C, D and E] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first (up to approximately 43 months)
  Duration of response (DoR), defined as the time from the first occurrence of a documented objective response to the time of the first documented disease progression per RECIST v1.1 or death from any cause, whichever occurs first
Preliminary anti-tumor activity of LUNA18 [Part A, AA, B, C, D and E] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first (up to approximately 43 months)
  Progression free survival (PFS), defined as the time from the first study treatment to the first occurrence of progression per RECIST v1.1 or death from any cause, whichever occurs first
Anti-drug antibody to LUNA18[Part A, AA, B, C, D and E] | From Cycle 0 Day 1 (Cycle 0 is 6-9 days) until study completion or treatment discontinuation (up to approximately 43 months)
  Incidence of anti-LUNA18 antibodies
Plasma concentrations of LUNA18 [Part B, C and E] | From Cycle 0 Day 1 (Cycle 0 is 6-9 days) until study completion or treatment discontinuation (up to approximately 43 months)
  Plasma concentrations of LUNA18
Phosphorylation level of ERK protein (pERK) in tumor tissues [Part A, AA, C, D, E] | From screening until the time of clinical responses and/or the time of progressive disease (up to approximately 43 months), if feasible
  Phosphorylation level of ERK protein (pERK) in tumor tissues biomarkers as applicable in tumor tissues

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (20):
- United States (13):
  - University of California - Davis, Davis, California
  - Beth Israel Deaconess, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - Renown Regional Medical Center, Reno, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital-Comprehensive Cancer Center, Providence, Rhode Island
  - NEXT Oncology, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia
  - University of Wisconsin - Carbone Cancer Center, Madison, Wisconsin
- Japan (7):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Osaka International Cancer Institute, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).